CLINICAL TRIAL: NCT00241371
Title: A Phase II Study of Clofarabine in Patients With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No response seen in patients
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-0916
Record Dates: First submitted 2005-10-17; First posted 2005-10-18 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Clofarabine

ARMS (1):
- Clofarabine (Experimental): 4 mg/m2 IV over 1 hour on days 1-5 of each 28 day cycle.
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine

SUMMARY:
To determine the overall response rate (CR+PR) of patients with relapsed or refractory multiple myeloma treated with clofarabine.

DETAILED DESCRIPTION:
To determine the time to response, duration of response, and time to progression of patients treated with clofarabine.

To determine the safety and tolerability of clofarabine in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Multiple myeloma diagnosed by standard criteria.
2. Measurable levels of monoclonal protein in serum (>= 0.5 g/dL) or urine (>= 0.2 g/24 hr).
3. At least 1 prior therapies for multiple myeloma with documented evidence of progression on the most recent treatment.
4. Age 18 years or older.
5. ECOG performance status <= 2.
6. Acceptable organ and marrow function as defined below:

   * Hemoglobin >= 8 gm/dL
   * Absolute neutrophil count >= 1,000/mm3
   * Platelets >= 50,000/mm3
   * Total bilirubin <= 2.5 X institutional upper limit of normal
   * AST, ALT <= 2.5 X institutional upper limit of normal
   * Creatinine 1.5 x institutional upper limit of normal
   * Normal cardiac function as determined by standard institutional methods
7. Women of child bearing potential must agree to use adequate contraception prior to study entry and for the duration of study.
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Receiving any other investigational agents.
2. Receiving concurrent steroids with a dose equivalent of prednisone of >= 150 mg/month.
3. Pregnant or nursing.
4. Active systemic infection considered opportunistic, life threatening or clinically significant at the time of treatment.
5. Severe concurrent disease, including severe insulin-dependent diabetes, uncontrolled hypertension, transient ischemic attacks, uncontrolled symptomatic coronary artery disease, or symptomatic CNS involvement or psychiatric illness/social situations that would limit compliance with study requirements.
6. History of other malignancy except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast unless the subject has been off treatment and free from disease for >= 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-03; Primary Completion 2005-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Overall response rate (CR+PR) | Every 3 months

SECONDARY OUTCOMES:
Time to response | Every 3 months
Safety and tolerability of clofarabine | 30 days after last treatment
Duration of response | Every 3 months
Time to progression | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Vij, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu